CLINICAL TRIAL: NCT02855645
Title: The Effects of Trichosanthes Root on Blood Sugar in Patients With Diabetes Mellitus
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH105-REC2-052
Record Dates: First submitted 2016-07-21; First posted 2016-08-04 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus
Keywords: Trichosanthes root; Traditional Chinese Medicine; Clinical trial
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Trichosanthes root (Experimental): Trichosanthes root at a rate of 1.5 g two times per day for 84 days.
  Interventions: Drug: Trichosanthes root
- Placebo (Placebo Comparator): Trichosanthes root at a rate of 0.15g (10%) two times per day for 84 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trichosanthes root — Trichosanthes root at a rate of 1.5 g two times per day for 84 days.
  Arms: Trichosanthes root
Drug: Placebo — Trichosanthes root at a rate of 0.15g (10%) two times per day for 84 days.
  Arms: Placebo

SUMMARY:
Diabetes mellitus (DM) locates fifth of ten leading death etiology, the population of diabetic patients has a tendency of increase. Trichosanthes root is called as Tian Hua Fen, According to traditional Chinese writing record that Trichosanthes root has the action of downbear fire, moisten dryness, and slippery phlegm, and release thirst. The Trichosanthes root may lower blood sugar levels in the modern study. The investigators designed a double blind, randomized controlled study, a total of 60 diabetic patients with high blood sugar were divided into treatment and control groups, and each group was 30 patients. In the treatment group, oral administration of Trichosanthes root 1.5 g, bid/day for 84 days continuously; in the control group, oral administration of Trichosanthes root placebo 1.5 g, bid/day for 84 days continuously. The main outcome measure was the changes of plasma blood sugar and Glycated hemoglobin A1c (HbA1c) levels changed before and after Trichosanthes root treatment. The investigators predict the results of the present study indicated that Trichosanthes root can improve plasma blood sugar and glycated hemoglobin A1c levels.

ELIGIBILITY:
Inclusion Criteria:

1. Early diagnosis Type Ⅱ Diabetic patients who Glycated hemoglobin A1c level between 7.0% and 9.0% (including) , and after three months of diet and exercise control.
2. The subject who was taking hypoglycemic drugs Metformin, the maximum total amount of ≦ 1500 mg / day.
3. Age ranged between 20 and 80 years (including).

Exclusion Criteria:

1. Pregnancy or breast-finding.
2. Allergy to test medicine.
3. Type I Diabetic patients.
4. Bleeding tendency.
5. The participants who suffered from serious disorders, such as congestive heart failure, myocardial infarction, chronic obstructive pulmonary disease, renal failure, cancer or stroke etc.
6. Irritable or anxious patients who cannot be assessed.
7. Refuse to sign the agreement.
8. The values of SGOT and SGPT levels were more than normal limit triple, or the value of creatinine level was more than normal limit.
9. Plasm glucose(Glucose AC) level in fasting state ≧ 300 mg / dL.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin A1c | Three months
  Improvement of glycated hemoglobin A1c levels
Plasma Blood Sugar | Three months
  Improvement of Plasma Blood Sugar levels

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Liang Hsieh, Study Chair — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan